CLINICAL TRIAL: NCT05745220
Title: Corneal Sensitivity in Silicone Hydrogel Contact Lens Wear
Brief Title: Influence of Silicone Hydrogel Contact Lens Neophyte Wear on Corneal Sensitivity
Acronym: CSCL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Daniela Nosch (Other)
Responsible Party: Sponsor-Investigator, Daniela Nosch, Clinical Professor, University of Applied Sciences and Arts Northwestern Switzerland
Organization: University of Applied Sciences and Arts Northwestern Switzerland (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2022-D0124
Record Dates: First submitted 2023-02-16; First posted 2023-02-27 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Cornea
Keywords: silicone hydrogel contact lens; daily contact lens wear; corneal sensitivity; esthesiometry
MeSH Terms: conditions — Corneal Diseases

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Daily contact lens wear (Other): Participant wear silicone hydrogel contact lenses daily for 6 weeks ±2 days for a minimum wearing time of 5 days per week and 8 hours per day - corneal sensitivity will be measured and compared at baseline versus after 7±2 days and 5 weeks ±2 days daily contact lens wear.
  Interventions: Other: Device: silicone hydrogel contact lens

INTERVENTIONS:
Other: Device: silicone hydrogel contact lens — Silicone hydrogel contact lens

SUMMARY:
Soft contact lenses can affect the ocular surface and sometimes cause intolerance. The aim of this study is to measure corneal sensitivity using the Swiss Liquid Jet aesthesiometer at baseline, after one and after six weeks, in novice daily contact lens wearers.

DETAILED DESCRIPTION:
Contact lens discomfort is described by many wearers. Wearing contact lenses can influence corneal sensitivity through three mechanisms: hypoxic, mechanical and inflammatory. A change in corneal sensitivity can be considered an indicator of a change in corneal physiology. Corneal sensitivity plays a major role in maintaining eye health. The interest of this study is to test the variability of the corneal sensitivity threshold during a new adaptation of silicone hydrogel contact lenses, and to verify whether there is a correlation with the wearer's comfort. For that, corneal sensitivity threshold measurements are taken at the baseline and then after one and six weeks of daily contact lens wear. The measurement is performed with the Swiss Liquid Jet aesthesiometer for corneal sensitivity (SLACS). After one week and six weeks of daily lens wear, participants complete a Contact Lens Dry Eye Questionnaire (CLDEQ-8) for comfort analysis.

ELIGIBILITY:
Inclusion Criteria:

* The Ocular Surface Disease Index questionnaire (OSDI) score for dry eye classification is ≤ 13
* Participants must be candidates for contact lens wear.
* Corneal radius between 7.4mm and 8.0mm
* If the corneal radius is > 8.0mm, the corneal diameter must be greater than 12.0mm.
* If the corneal radius is <7.4mm, the required corneal diameter is less than 12.0mm.
* Participants have a CL cylindrical ametropia ≤ -1.25 D.
* Participants will not have worn CL for 7 days prior to the start of the study.
* Participants do not wear CL regularly (no more than 1 days per week) prior to the start of the study.
* During the study, the participant wore the CL a minimum of 5 days per week for a minimum of 8 hours.
* The person being tested is in good health. This means that he or she does not suffer from any systemic diseases, such as diabetes or rheumatism, which could have an influence on eye health. He or she also has no eye disease and has not previously undergone corneal (refractive) surgery.

Exclusion Criteria:

* The participant is a minor.
* The participant has worn CL within the last 7 days.
* The radius of the cornea is not within the prescribed range. In addition, the corneal diameter is not within the prescribed range either.
* The participant's ametropia is not within the prescribed range.
* The participant has worn the lenses for less than 8 hours for less than five days.
* The participant has no diagnosis of dry eye.
* The OSDI questionnaire score for the Dry Eye classification is greater than 13.
* The participant suffers from a systemic disease (diabetes or rheumatism) that could influence ocular health, an ocular disease or has already undergone refractive surgery.
* Vulnerable participants

Ages: 18 Years to 38 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2023-04-08 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Difference in corneal sensitivity threshold baseline and after one and six weeks of daily contact lens wear | 7±2 days and 5 weeks ±2
  Comparison of corneal sensitivity threshold at the baseline and after one and six weeks of daily wear of silicone hydrogel contact lenses on neophyte wearer. Corneal sensitivity measurement will take place with the Swiss Liquid Jet Aesthesiometer for Corneal Sensitivity (SLACS) and will be recorded in mbar.

SECONDARY OUTCOMES:
Correlation between corneal sensitivity threshold and subjective symptoms | 7±2 days and 5 weeks ±2
  Correlation between corneal sensitivity threshold and subjective symptoms after one and six weeks of daily contact lens wear: corneal sensitivity threshold will be determined with the Swiss Liquid Jet Aesthesiometer for Corneal Sensitivity (SLACS) and will be recorded in mbar. Subjective Symptoms will be recorded with the Contact Lens Dry Eye Questionnaire (CLDEQ-8) scored from 0=comfortable to 37=uncomfortable (specifically designed to assess contact lens comfort)

CONTACTS AND LOCATIONS:
Overall Officials: Daniela Nosch, PhD, Principal Investigator — Institute of Optometry, FHNW
Locations (1):
- Optique Messerli Optometry centre, Marly, Canton of Fribourg, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Belmonte C, Acosta MC, Gallar J. Neural basis of sensation in intact and injured corneas. Exp Eye Res. 2004 Mar;78(3):513-25. doi: 10.1016/j.exer.2003.09.023. PMID 15106930
- [Background] Morgan PB, Murphy PJ, Gifford KL, Gifford P, Golebiowski B, Johnson L, Makrynioti D, Moezzi AM, Moody K, Navascues-Cornago M, Schweizer H, Swiderska K, Young G, Willcox M. CLEAR - Effect of contact lens materials and designs on the anatomy and physiology of the eye. Cont Lens Anterior Eye. 2021 Apr;44(2):192-219. doi: 10.1016/j.clae.2021.02.006. Epub 2021 Mar 25. PMID 33775377
- [Background] Muller LJ, Marfurt CF, Kruse F, Tervo TM. Corneal nerves: structure, contents and function. Exp Eye Res. 2003 May;76(5):521-42. doi: 10.1016/s0014-4835(03)00050-2. PMID 12697417
- [Background] Nosch DS, Oscity M, Steigmeier P, Kaser E, Loepfe M, Joos RE. Working principle and relevant physical properties of the Swiss Liquid Jet Aesthesiometer for Corneal Sensitivity (SLACS) evaluation. Ophthalmic Physiol Opt. 2022 May;42(3):609-618. doi: 10.1111/opo.12962. Epub 2022 Feb 14. PMID 35156726
- [Background] Stapleton F, Marfurt C, Golebiowski B, Rosenblatt M, Bereiter D, Begley C, Dartt D, Gallar J, Belmonte C, Hamrah P, Willcox M; TFOS International Workshop on Contact Lens Discomfort. The TFOS International Workshop on Contact Lens Discomfort: report of the subcommittee on neurobiology. Invest Ophthalmol Vis Sci. 2013 Oct 18;54(11):TFOS71-97. doi: 10.1167/iovs.13-13226. PMID 24058137
- [Background] Nichols JJ, Willcox MD, Bron AJ, Belmonte C, Ciolino JB, Craig JP, Dogru M, Foulks GN, Jones L, Nelson JD, Nichols KK, Purslow C, Schaumberg DA, Stapleton F, Sullivan DA; members of the TFOS International Workshop on Contact Lens Discomfort. The TFOS International Workshop on Contact Lens Discomfort: executive summary. Invest Ophthalmol Vis Sci. 2013 Oct 18;54(11):TFOS7-TFOS13. doi: 10.1167/iovs.13-13212. No abstract available. PMID 24058135